CLINICAL TRIAL: NCT01405287
Title: A Prospective Randomized Study to Compare Vascular Healing After Deployment of the Abluminal Sirolimus Coated Bio-Engineered (Combo) Stent Versus the Everolimus Eluting Stent in Patients With Acute Coronary Syndrome by Means of OCT
Brief Title: Study of Vascular Healing With the Combo Stent Versus the Everolimus Eluting Stent in ACS Patients by Means of OCT
Acronym: REMEDEE-OCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OrbusNeich (Industry)
Collaborators: Genae (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VP-0509; 36383 (Other: CCMO)
Record Dates: First submitted 2011-07-26; First posted 2011-07-29 (Estimated); Last update posted 2014-03-24 (Estimated); Status verified 2014-03

CONDITIONS: Coronary Artery Disease; Atherosclerosis; Acute Coronary Syndrome (ACS); Myocardial Infarction (MI)
Keywords: stent; drug eluting stent; healing; endothelium; DES; OCT; MI; ACS
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis; Acute Coronary Syndrome; Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Combo Stent (Experimental): PTCA with Combo Stent
  Interventions: Device: PTCA with stent placement
- Everolimus Eluting Stent (EES) (Active Comparator): PTCA with DES (Everolimus Eluting Stent: Xience V or Promus)
  Interventions: Device: PTCA with stent placement

INTERVENTIONS:
Device: PTCA with stent placement — PTCA with stent placement (Drug Eluting Stent)
  Other Names: Combo Stent; Xience V or Promus stent

SUMMARY:
OBJECTIVE It is the objective of the REMEDEE OCT study to assess vascular healing after deployment of the Abluminal Sirolimus Coated Bio-Engineered Stent (Combo Bio-Engineered Sirolimus Eluting Stent) in patients with Acute Coronary Syndrome (ACS) with single de novo native coronary artery lesions ranging in diameter from ≥2.5 mm to ≤3.5 mm and ≤ 20 mm in length.

STUDY DESIGN The REMEDEE OCT study is a prospective, multicenter, randomized study designed to enroll 60 patients with ACS who will be randomized 1:1 to be treated with the Combo stent versus the commercially available everolimus eluting stent (Xience V or Promus). Patients will receive Optical Coherence Tomography (OCT) and Quatitative Coronary Angiography (QCA) follow-up imaging at 60 days post procedure. Clinical follow-up is scheduled at 30, 60, 180, 360 and 540 days. Furthermore, QCA and OCT will also be performed at baseline in all participants of the study.

DETAILED DESCRIPTION:
BACKGROUND The implantation of bare-metal stents (BMS) has significantly reduced clinical and angiographic restenosis compared to balloon angioplasty alone after PCI due to eliminating elastic recoil and reducing arterial remodeling. However, in-stent restenosis still occurred frequently after BMS implantation in 20% to 40% of patients due to neointimal proliferation. The development, clinical validation and widespread use of drug-eluting stents (DES) have revolutionized the treatment of patients with coronary artery disease. Large-scale, prospective, multicenter double-blind randomized trials have provided strong evidence that drug-eluting stents significantly reduce angiographic restenosis and enhance event-free survival compared with BMS after implantation in native coronary arteries (3-6).However, despite an improved efficacy in the prevention of restenosis and target vessel failure safety concerns have been raised for DES, focusing on a small but clinically important increase in stent thrombosis occurring greater than one year after the index procedure.

In patients receiving drug-eluting stents, the acute coronary syndrome has been identified as one of the major risk factors of stent thrombosis (10). Therefore, concerns about the long-term outcome and safety after drug-eluting stent implantation due to late stent thrombosis and late stent malapposition have been raised.

Stent thrombosis, in particular late stent thrombosis, has been related to an impaired stent healing, most of all to a reduced endothelial repair, i.e. reduced stent strut coverage, after implantation of drug-eluting stents. This has resulted in the recommendation of a prolonged 12-month double antiplatelet therapy with aspirin and clopidogrel after drug-eluting stent implantation, however, how long double antiplatelet therapy is needed is unknown at present. These observations have resulted in an intense search for alternative strategies to promote stent healing and endothelial repair, rather than to inhibit the endothelialisation of the stent, that is common to the substances used to prevent neointima formation.

Notably, endothelial repair can be substantially stimulated by CD34+ endothelial progenitor cells. The Combo stent is therefore covered with a CD34+ antibody to attract endothelial progenitor cells to promote endothelial and stent healing, and on the abluminal side releases sirolimus to prevent neointima formation and restenosis. Several preclinical studies in the porcine coronary artery model have shown, that endothelialisation and stent healing are accelerated in the Combo stent. The present study has therefore been designed to compare stent healing of the Combo stent with the everolimus-eluting stent by optical coherence tomography analysis (optical frequency domain imaging; OFDI), a high resolution intracoronary imaging technique allowing accurate evaluation of stent coverage and healing, in patients with an acute coronary syndrome. Previous studies have indicated, that coronary stent healing after DES implantation is particularly impaired in patients with ACS, and therefore this patient population is in a particular need of improved "pro-healing" stent concepts with a high efficacy.

RATIONALE An important limitation of stents eluting only growth-inhibiting substances is, that also the desirable endothelial cell growth over the stent struts is prevented, that is thought to represent a major cause of "late-stent-thrombosis". The rationale for the design of the "combo-stent" is therefore to combine a growth inhibiting substance with abluminal release with an endothelial progenitor cell attracting design to promote endothelial repair. In the pre-clinical studies, the "Combo Stent" demonstrated significantly lower neointimal hyperplasia, while also showing improved endothelial coverage relative to other commercially available DES. There was also a noticeably lower presence of inflammation and foreign body reaction.

OCT- Examination of Vessel Healing Optical coherence tomography (OCT) is a novel intravascular imaging modality based on infrared light emission that has a 10-20 fold higher resolution (10-20 µM) as compared to current intravascular ultrasound systems, and allows a detailed examination of stent healing. Strut coverage, strut apposition and neointima can be quantified at a micron-scale level with a resolution 10-20 times higher than conventional intravascular ultrasound. The quantification of stent healing by intravascular OCT analysis has recently been validated against histology, demonstrating an excellent accuracy of the OCT examination. Moreover, the safety and feasibility of OCT examination in a multicenter study has been demonstrated. Newer modalities of OCT image acquisition, as used in this study, have been reported to further simplify the technique and reduce procedural time.

ELIGIBILITY:
Inclusion Criteria

1. age ≥18 and ≤ 80 years
2. ST or Non-ST-segment elevation MI (assumed to be a type 1)
3. Acceptable CABG candidate
4. Patient willing to comply with specified follow-up
5. Patient or legally authorized representative has been informed of the nature of the study, agrees to its provisions and has been provided written informed consent
6. Single de novo or non-stented restenotic lesion in a native coronary artery
7. Patients with 2-vessel coronary disease, may have undergone successful treatment (<20% diameter stenosis by visual estimate) of the non-target vessel with approved devices up to and including the index procedure but must be prior to the index target vessel treatment. Any non-target vessel or lesion intended to be treated during the index procedure or follow-up, cannot be an unprotected left main, ostial lesion, chronic total occlusion, heavily calcified, bifurcation, vein grafts, be anything requiring atherectomy, thrombectomy, or pre-treatment with anything other than balloon angioplasty; 8. Target lesion (maximum length is 20 mm by visual estimate) to be covered by a single stent of max 23 mm (stent coverage incl at least 3 mm of healthy vessel is recommended). The lesion length to be measured after pre-dilation 9. Reference vessel diameter ≥2.5 to ≤ 3.5 mm by visual estimate 10. The vessel diameter should be measured after pre-dilation procedure and after intra-coronary nitroglycerin if spasm is suspected 11. Target lesion ≥50% and <100% stenosed by visual estimate

Exclusion Criteria

1. Pregnant or nursing patients and those who plan pregnancy in the period up to 1 year following index procedure. Female patients of childbearing potential must have a negative pregnancy test done within 7 days prior to the index procedure per site standard test
2. Impaired renal function or on dialysis
3. Platelet count <100,000 cells/mm3 or >700,000 cells/mm3 or a WBC<3,000 cells/mm3
4. Patient has a history of bleeding diathesis or coagulopathy or patients in whom anti-platelet and/or anticoagulant therapy is contraindicated
5. Patient requires low molecular weight heparin (LMWH) treatment postprocedure or has received a dose of LMWH ≤8 hours prior to index procedure
6. Patient has received any organ transplant or is on a waiting list for any organ transplant;
7. Patient has other medical illness or known history of substance abuse that may cause non-compliance with the protocol, confound the data interpretation or is associated with a limited life expectancy (<1 year)
8. Patient has a known hypersensitivity or contraindication to aspirin, heparin/bivalirudin, clopidogrel/ticlopidine, prasugrel, stainless steel alloy, sirolimus and/or contrast sensitivity that cannot be adequately pre-medicated
9. Patient has previously received murine therapeutic antibodies and exhibited sensitization through the production of Human Anti-Murine Antibodies
10. Patient presents with cardiogenic shock
11. Patient has extensive peripheral vascular disease that precludes safe 6 French sheath insertion;
12. Any significant medical condition which in the Investigator's opinion may interfere with the patient's optimal participation in the study
13. Currently participating in another investigational drug or device study or patient in inclusion in another investigational drug or device study during follow-up
14. Unprotected left main coronary artery disease with ≥50% stenosis
15. Ostial target lesion(s)
16. Totally occluded target vessel (TIMI flow 0)
17. Calcified target lesion(s) which cannot be successfully predilated
18. Target lesion has excessive tortuosity unsuitable for stent delivery and deployment;
19. Target lesion involving bifurcation with a side branch ≥2.0 mm in diameter (either stenosis of both main vessel and major side branch or stenosis of just major side branch) that would require intervention of diseased side branch
20. A significant (>50%) stenosis proximal or distal to the target lesion that cannot be covered by same single stent
21. Diffuse distal disease to target lesion with impaired runoff
22. Pre-treatment with devices other than balloon angioplasty
23. Prior stent within 10 mm of target lesion
24. Intervention (PCI or bypass) of any lesion in the target vessel performed within the previous 6 months
25. Intervention (PCI or bypass) of another lesion in a non-target vessel performed within 30 days prior to the index
26. Planned intervention of another lesion (target vessel or non-target vessel) within 30 days.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-10; Primary Completion 2012-08 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Percentage of uncovered stent struts per stent at follow-up (OCT) | 60 days

SECONDARY OUTCOMES:
Secondary Clinical Endpoint: Major Adverse Cardiac Events (MACE) | 30, 60, 180, 360, 540 days
  Major Adverse Cardiac Events (MACE)defined as a composite of death, Myocardial Infarction (MI) (Q wave or non-Q wave), emergent coronary artery bypass surgery (CABG), or justified target lesion revascularization (TLR) by repeat Percutaneous Transluminal Coronary Angioplasty (PTCA) or Coronary Artery Bypass Grafting (CABG) at hospital discharge
Secondary Clinical Endpoint: components of MACE: cardiac death | 30, 60, 180, 360, 540 days
  cardiac death
Secondary Clinical Endpoints: components of MACE: MI | 30, 60, 180, 360, 540 days
  MI (Q wave or non-Q wave)
Secondary Clinical Endpoints: components of MACE: CABG or re-PTCA of target lesion | 30, 60, 180, 360, 540 days
  emergent coronary artery bypass surgery (CABG), or clinically justified target lesion revascularization (TLR) by repeat PTCA or CABG at hospital discharge
Secondary Clinical Endpoints: Stent thrombosis | 30, 60, 180, 360, 540 days
  Target vessel stent thrombosis per Academic Research Consortium (ARC) definition
Secondary OCT Endpoints (1/12) | 60 days
  Percentage of stent strut malapposition
Secondary OCT Endpoints (2/12) | 60 days
  Maximum length of segments (mm) with uncovered struts
Secondary OCT Endpoints (3/12) | 60 days
  Maximum length of segments (mm) with malapposed struts
Secondary OCT Endpoints (4/12) | 60 days
  Maximum malapposition distance (mm)
Secondary OCT Endpoints (5/12) | 60 days
  Total malapposition volume
Secondary OCT Endpoints (6/12) | 60 days
  Maximal malapposition volume
Secondary OCT Endpoints (7/12) | 60 days
  Mean neointimal thickness (NIT)(strut level)
Secondary OCT Endpoints (8/12) | 60 days
  Percentage of protruding struts per stent
Secondary OCT Endpoints (9/12) | 60 days
  Frequency of Abnormal Intrastent Tissue (AIST)
Secondary OCT Endpoints (10/12) | 60 days
  Stent Volume
Secondary OCT Endpoints (11/12) | 60 days
  Lumen Volume
Secondary OCT Endpoints (12/12) | 60 days
  Neointimal Hyperplasia (NIH) Volume

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Landmesser, MD, PhD, Principal Investigator — University of Zurich
Locations (6):
- Belgium (2):
  - OLV Ziekenhuis Aalst, Aalst
  - AZ Middelheim, Antwerp
- Satakunta Central Hospital, Pori, Finland
- Academisch Medisch Centrum, Amsterdam, Netherlands
- University Hospital Zurich, Zurich, Switzerland
- King's College Hospital, London, United Kingdom

REFERENCES:
- [Derived] Jaguszewski M, Aloysius R, Wang W, Bezerra HG, Hill J, De Winter RJ, Karjalainen PP, Verheye S, Wijns W, Luscher TF, Joner M, Costa M, Landmesser U. The REMEDEE-OCT Study: An Evaluation of the Bioengineered COMBO Dual-Therapy CD34 Antibody-Covered Sirolimus-Eluting Coronary Stent Compared With a Cobalt-Chromium Everolimus-Eluting Stent in Patients With Acute Coronary Syndromes: Insights From Optical Coherence Tomography Imaging Analysis. JACC Cardiovasc Interv. 2017 Mar 13;10(5):489-499. doi: 10.1016/j.jcin.2016.11.040. PMID 28279316